CLINICAL TRIAL: NCT04415164
Title: A Multi-center, Randomized, Double-blind, Placebo-controlled Trial to Evaluate the Efficacy and Safety of Xueshuantong Lyophilized Powder in Chinese Patients With Acute Ischemic Stroke
Brief Title: Evaluation of Xueshuantong in Patients With AcutE IschemiC STroke
Acronym: EXPECT
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Dongzhimen Hospital, Beijing (Other)
Collaborators: Tianjin University of Traditional Chinese Medicine (Other)
Responsible Party: Principal Investigator, Ying Gao, President of Institute for Brain Disorders, Beijing University of Chinese Medicine, Dongzhimen Hospital, Beijing
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: P2019-08-BDY-08-V04
Record Dates: First submitted 2020-05-25; First posted 2020-06-04 (Actual); Last update posted 2021-04-09 (Actual); Status verified 2021-04

CONDITIONS: Acute Ischemic Stroke
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Xueshuantong (Experimental): Patients will receive intravenously administered Xueshuantong, combined with guidelines-based standard care.
  Interventions: Drug: Xueshuantong lyophilized powder; Other: Guidelines-based standard care
- Placebo (Placebo Comparator): Patients will receive intravenously administered Xueshuantong placebo, combined with guidelines-based standard care.
  Interventions: Drug: Placebo; Other: Guidelines-based standard care

INTERVENTIONS:
Drug: Xueshuantong lyophilized powder — Xueshuantong lyophilized powder (500mg), diluted with 250 ml of 0.9% sodium chloride injection, IV (in the vein), once a day, continue for 10 days.
  Other Names: Zhusheyong Xueshuantong (donggan); WS-10460(ZD-0460)-2002-2011Z
  Arms: Xueshuantong
Drug: Placebo — Xueshuantong lyophilized powder Placebo. The usage of placebo is the same as that in the experimental group.
  Arms: Placebo
Other: Guidelines-based standard care — Guidelines-based standard care for acute ischemic stroke

SUMMARY:
The aim is to assess the effects and harms of Xueshuantong lyophilized powder versus placebo in patients with acute ischemic stroke when initiated within 72 hours of symptom onset.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of acute ischemic stroke.
2. Patients that can be treated with study drug within 72 hours of symptoms onset defined by the "last see normal" principle.
3. 4 ≤ NIHSS score ≤ 16 (total score of upper and lower limbs on motor deficits ≥ 2) at the randomization time.
4. Female or male aged ≥ 18 years and ≤ 80 years.
5. Provision of signed informed consent prior to any study-specific procedure.

Exclusion Criteria:

1. Patients who have received intravenous/intra-arterial thrombolysis or mechanical thrombectomy prior to randomization.
2. Secondary stroke caused by tumor, traumatic brain Injury, hematological disease or other diseases with the explicit diagnosis.
3. mRS grade ≥ 2 pre-morbid historical assessment.
4. Other conditions that lead to motor dysfunction (e.g. claudication, severe osteoarthrosis, rheumatoid arthritis, gouty arthritis or other diseases).
5. Known severe impairment of liver function or renal function.
6. Known hypersensitivity to study drugs.
7. Known severe comorbidity with life expectancy < 3 months.
8. Known massive cerebral infarction combined with disturbance of consciousness (1a ≥ 2 in NIHSS), dementia, mental impairment, or unsuitable for participation, in the opinion of the investigator.
9. Pregnancy or breastfeeding.
10. Participation in another clinical study with an investigational product at any time during the 3 months prior to randomization (regardless of when treatment with the investigational product was discontinued).

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 480 (Estimated)
Dates: Start 2020-09-29 (Actual); Primary Completion 2022-10-31 (Estimated); Study Completion 2023-05-31 (Estimated)

PRIMARY OUTCOMES:
Change in National Institute of Health Stroke Scale score on day 10 (after the treatment) from baseline | Day 10 ± 2
  The aim is to assess the effects of Xueshuantong lyophilized powder versus placebo on reducing the neurological impairment when initiated within 72 hours of symptom onset in patients with acute ischemic stroke.
  The National Institute of Health Stroke Scale is a tool used by healthcare providers to objectively quantify the impairment caused by a stroke. It is composed of 11 items, each of which scores a specific ability between a 0 and 4. For each item, a score of 0 typically indicates normal function in that specific ability, while a higher score is indicative of some level of impairment. The individual scores from each item are summed in order to calculate a patient's total NIHSS score. The maximum possible score is 42, with the minimum score being a 0.

SECONDARY OUTCOMES:
The proportion of patients with National Institute of Health Stroke Scale score 0-1 on day 10 (after the treatment) | Day 10 ± 2
  The National Institute of Health Stroke Scale is a tool used by healthcare providers to objectively quantify the impairment caused by a stroke. It is composed of 11 items, each of which scores a specific ability between a 0 and 4. For each item, a score of 0 typically indicates normal function in that specific ability, while a higher score is indicative of some level of impairment. The individual scores from each item are summed in order to calculate a patient's total NIHSS score. The maximum possible score is 42, with the minimum score being a 0.
Patients-reported outcome of patients measured by Patient-Reported Outcomes Scale for Stroke on day 10 (after the treatment) | Day 10 ± 2
  Patient-Reported Outcomes Scale for Stroke, a structured questionnaire-scale was developed suitable for Chinese patients. The score ranges from 0 (best) to 144 (worst).
The proportion of patients with modified Rankin Scale grade ≤1 on day 90 | Day 90 ± 7
  Modified Rankin Scale, a commonly used scale for measuring the degree of dependence in the daily activities of people who have suffered a stroke or other causes of neurological disability. 0 - No symptoms.1 - No significant disability. Able to carry out all usual activities, despite some symptoms.2 - Slight disability. Able to look after own affairs without assistance, but unable to carry out all previous activities.3 - Moderate disability. Requires some help, but able to walk unassisted.4 - Moderately severe disability. Unable to attend to own bodily needs without assistance, and unable to walk unassisted.5 - Severe disability. Requires constant nursing care and attention, bedridden, incontinent.6 - Dead. The mRS grade between 3 to 6 points are considered to be poor functional outcome.
The proportion of patients with Barthel Index (BI) score greater than or equal to 90 on day 90 | Day 90 ± 7
  Barthel Index is a commonly used scale for measuring the activity of daily living of people. Score of 10-item scale ranges from 0 (worst) to 100 (best).
Quality of life of patients measured by Stroke-specific quality of life scale on day 90 | Day 90 ± 7
  Stroke-Specific Quality of Life Scale is a standardized instrument for evaluating health-related quality of life. The score of 49-item scale with 12 domains range from 49 (worst) to 245 (best).
Incidence of treatment-related adverse events | Up to Day 90
  Number of patients with any adverse events during the study.

OTHER OUTCOMES:
Change in intercellular adhesion molecule 1 level on day 10 (after the treatment) from baseline | Day 10 ± 2
  Level of intercellular adhesion molecule 1 is associated with the clinical outcome.
Change in Interleukin 6 level on day 10 (after the treatment) from baseline | Day 10 ± 2
  Level of Interleukin 6 is associated with the clinical outcome.
Change in tumor necrosis factor-α level on day 10 (after the treatment) from baseline | Day 10 ± 2
  Level of tumor necrosis factor-α is associated with the clinical outcome.
Change in matrix metalloproteinase 9 level on day 10 (after the treatment) from baseline | Day 10 ± 2
  Level of matrix metalloproteinase 9 is associated with the clinical outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Ying Gao, Principal Investigator — Dongzhimen Hospital, Beijing
Locations (1):
- Dongzhimen Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No